CLINICAL TRIAL: NCT00008125
Title: Phase I Study Of Gemcitabine, Docetaxel And Carboplatin, With And Without Filrastim Support, Combination Chemotherapy In Patients With Advanced Non-Hematological Malignancies
Brief Title: Combination Chemotherapy With or Without Filgrastim in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: PCI-97-093; CDR0000068377 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-980207; NCI-G00-1884
Record Dates: First submitted 2001-01-06; First posted 2004-05-04 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Filgrastim; Carboplatin; Docetaxel; Gemcitabine

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of gemcitabine combined with docetaxel and carboplatin with or without filgrastim in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of gemcitabine and docetaxel when administered with carboplatin with or without filgrastim (G-CSF) in patients with advanced solid tumors. II. Determine a safe dose level and schedule for this regimen for phase II study in these patients. III. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of docetaxel and gemcitabine. Patients receive gemcitabine IV over 30 minutes, docetaxel IV over 1 hour, and carboplatin IV over 30 minutes on day 1. Patients also receive gemcitabine IV over 30 minutes on day 8. Treatment repeats every 21 days for approximately 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of gemcitabine and docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). If the DLT is grade 4 neutropenia, filgrastim (G-CSF) is added to the regimen (administered subcutaneously on days 2-7 and 8-14 or until blood counts recover). A new MTD is then determined. Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed solid tumor for which no curative therapy exists No symptomatic or uncontrolled brain or leptomeningeal metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST no greater than 1.5 times ULN Renal: Creatinine no greater than ULN Cardiovascular: No unstable cardiac disease requiring treatment No new onset crescendo or rest angina Stable exertion angina allowed Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use 2 methods of contraception for at least 1 week prior to study, during study, and for at least 2 weeks after study No symptomatic peripheral neuropathy greater than grade 1 No significant neurologic or psychiatric disorders including psychotic disorders, dementia, or seizures No other significant medical or psychiatric condition that would preclude study No active infection No other malignancy within past 5 years except non-melanoma skin cancer, carcinoma in situ of the cervix, or other cancer that, due to its stage, is highly unlikely to recur during treatment No known hypersensitivity to E. coli-derived products

PRIOR CONCURRENT THERAPY: Biologic therapy: No other concurrent prophylactic hematopoietic growth factors (i.e., filgrastim (G-CSF) or sargramostim (GM-CSF)) Chemotherapy: No more than 1 prior chemotherapy regimen for advanced disease At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered Prior cisplatin, carboplatin, docetaxel, paclitaxel, or gemcitabine allowed No other concurrent chemotherapy Endocrine therapy: At least 3 weeks since prior hormonal therapy and recovered Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified Other: At least 3 weeks since prior investigational drugs and recovered No other concurrent experimental agents No other concurrent anti-cancer therapy No concurrent prophylactic oral or IV antibiotics without fever present

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1998-03; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P. Belani, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States